CLINICAL TRIAL: NCT00005849
Title: Phase II Study of Bryostatin-1 in Combination With Paclitaxel for Non-Small Cell Lung Cancer
Brief Title: Bryostatin 1 Plus Paclitaxel in Treating Patients With Stage IIIB, Stage IV, or Recurrent Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10337; UCCRC-10337; NCI-T99-0018
Record Dates: First submitted 2000-06-02; First posted 2004-04-26 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — bryostatin 1; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental): Paclitaxel (90 mg/m2, days 1, 8 and 15 of every 28 day cycle), Bryostatin-1 (50 mcg/m2, days 2, 9 and 16 of every 28 day cycle)
  Interventions: Drug: bryostatin 1; Drug: paclitaxel

INTERVENTIONS:
Drug: bryostatin 1
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of bryostatin 1 plus paclitaxel in treating patients who have stage IIIB, stage IV, or recurrent non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the overall, partial, and complete response rates in patients with stage IIIB-IV or recurrent non-small cell lung cancer treated with bryostatin 1 and paclitaxel. II. Determine the overall survival and time to tumor progression in patients treated with this regimen. III. Determine the T cell subset analysis and serum levels of interleukin-6 and tumor necrosis factor alpha in these patients after receiving bryostatin 1 and correlate with clinical endpoints.

OUTLINE: This is a multicenter study. Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15 and bryostatin 1 IV over 1 hour on days 2, 9, and 16. Treatment repeats every 4 weeks for a minimum of 2 courses in the absence of disease progression or unacceptable toxicity. Patients are followed for at least 2 years for survival.

PROJECTED ACCRUAL: A total of 15-40 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven stage IIIB, IV or recurrent non-small cell lung cancer (NSCLC) Patients with stage IIIB disease must have pleural effusion Measurable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Karnofsky 50-100% Life expectancy: Not specified Hematopoietic: WBC greater than 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin normal SGOT less than 2 times normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 50 mL/min Blood urea nitrogen less than 1.5 times normal Cardiovascular: No symptomatic congestive heart failure, unstable angina pectoris, or myocardial infarction within the past 6 months No heart block worse than first degree, bundle branch block, or ventricular or supraventricular arrhythmia by 12 lead electrocardiogram Other: Not pregnant or nursing Fertile patients must use effective contraception No uncontrolled concurrent illness including, but not limited to, ongoing or active infection

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent colony-stimulating factors Chemotherapy: No prior chemotherapy for NSCLC Endocrine therapy: Not specified Radiotherapy: Greater than 4 weeks since prior radiotherapy Surgery: Not specified Other: No other concurrent investigational agents No concurrent antiretroviral therapy (HAART) in HIV positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2000-04; Primary Completion 2002-09 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Clinical response rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ann M. Mauer, MD, Study Chair — University of Chicago
Locations (10):
- United States (10):
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Evanston Northwestern Health Care, Evanston, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Michiana Hematology/Oncology P.C., South Bend, Indiana

REFERENCES:
- [Result] Winegarden JD, Mauer AM, Gajewski TF, Hoffman PC, Krauss S, Rudin CM, Vokes EE. A phase II study of bryostatin-1 and paclitaxel in patients with advanced non-small cell lung cancer. Lung Cancer. 2003 Feb;39(2):191-6. doi: 10.1016/s0169-5002(02)00447-6. PMID 12581572